CLINICAL TRIAL: NCT01759303
Title: A Phase II Study of Pazopanib in the Treatment of Osteosarcoma Metastatic to the Lung
Brief Title: Study of Pazopanib in the Treatment of Osteosarcoma Metastatic to the Lung
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: low accrual
Sponsor: Emerald Clinical Inc. (Industry)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AWACMOS1102
Record Dates: First submitted 2012-12-21; First posted 2013-01-03 (Estimated); Last update posted 2021-04-13 (Actual); Status verified 2021-04

CONDITIONS: Osteosarcoma; Metastatic Osteosarcoma
MeSH Terms: conditions — Osteosarcoma | interventions — pazopanib

STUDY DESIGN:
Masking Description: Open Label
Oversight: Data Monitoring Committee: No

ARMS (1):
- pazopanib (Experimental): For subjects > 18 years of age and subjects 16-17 years of age with a BSA ≥ 1.6 Pazopanib 800mg once daily will be started on Cycle 1 Day 1 and will be administered continuously for each 28-day cycle. Subjects may continue study treatment until they develop disease progression or unacceptable toxicity.
  For subjects 16-17 years of age with a BSA < 1.6 m2, Pazopanib 600mg once daily will be started on Cycle 1 Day 1 and will be administered continuously for each 28-day cycle. Subjects may continue study treatment until they develop disease progression or unacceptable toxicity.
  Interventions: Drug: pazopanib

INTERVENTIONS:
Drug: pazopanib — For subjects > 18 years of age and subjects 16-17 years of age with a BSA ≥ 1.6 Pazopanib 800mg once daily will be started on Cycle 1 Day 1 and will be administered continuously for each 28-day cycle. Subjects may continue study treatment until they develop disease progression or unacceptable toxicity.
  For subjects 16-17 years of age with a BSA < 1.6 m2, Pazopanib 600mg once daily will be started on Cycle 1 Day 1 and will be administered continuously for each 28-day cycle. Subjects may continue study treatment until they develop disease progression or unacceptable toxicity.
  Other Names: Votrient

SUMMARY:
The purpose of this study is to determine the 4-month Progression-Free Survival (PFS), with demonstrated increase in tumor doubling time, of eligible subjects treated with pazopanib according to RECIST version 1.1 guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent or assent
* Age > or = to 16 years
* Histologically confirmed diagnosis of osteosarcoma with lung metastasis, who have progressed on the prior line of therapy, or relapsed
* Ineligible for curative pulmonary metastasectomy
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 guidelines. At least one measurable lesion must be in the lungs.
* Eligible subjects are required to have > or = to 1 line of multi-agent chemotherapy either neoadjuvantly or adjuvantly. Subjects may have had 0-2 lines of therapy for metastatic disease.
* Measured cardiac ejection fraction > or = to 50% or the institutional lower limit of normal by echocardiogram or MUGA scan.
* Adequate organ system function.
* Females must be either non-child bearing potential or have a negative pregnancy test within 3 to 5 days prior to the first dose of study drug.

Exclusion Criteria:

* Children not in the care or custody of a biological parent, adoptive parent, appointed legal guardian, or legally appointed foster care.
* Prior exposure to VEGFR tyrosine kinase inhibitor (small molecule or antibody) or VEGFR antibody.
* Prior malignancy. Note: Subjects who have had another malignancy and have been disease-free for 3 years, or subjects with a history of completely resected non-melanomatous skin carcinoma or successfully treated in situ carcinoma are eligible.
* History or clinical evidence of central nervous system (CNS) metastases or leptomeningeal carcinomatosis, unless previously treated, asymptomatic, and off steroids and anti-seizure medication for 6 months prior to first dose of study drug
* Clinically significant gastrointestinal abnormalities that may increase the risk for gastrointestinal bleeding.
* Clinically significant gastrointestinal abnormalities that may affect absorption of investigational product.
* Presence of uncontrolled infection.
* Corrected QT interval (QTc) > 480 msecs using Bazett's formula.
* History of certain cardiovascular conditions within the past 6 months.
* Class II-IV congestive heart failure, as defined by the New York Heart Association
* Poorly controlled hypertension [defined as systolic blood pressure (SBP) of ≥ 140 mmHg or diastolic blood pressure (DBP) of ≥ 90mmHg].
* History of cerebrovascular accident including transient ischemic attack (TIA), pulmonary embolism or untreated deep venous thrombosis (DVT) within the past 6 months.
* Prior major surgery or trauma within 28 days prior to the protocol-mandated 4-week drug holiday and/or presence of any non-healing wound, fracture, or ulcer.
* Evidence of active bleeding or bleeding diathesis.
* Known endobronchial lesions and/or lesions infiltrating major pulmonary vessels that increase the risk of pulmonary hemorrhage.
* Hemoptysis of red blood in excess of 2.5 mL (or one half teaspoon) within 8 weeks of first dose of study drug.
* Any serious and/or unstable pre-existing medical, psychiatric, or other condition that could interfere with subject's safety, provision of informed consent/assent, or compliance to study procedures.
* Unable or unwilling to discontinue use of prohibited medications for at least 14 days or five half-lives of a drug, whichever is longer, prior to the first dose of study drug and for the duration of the study treatment.
* Radiation therapy, minor surgery, tumor embolization, chemotherapy, immunotherapy, biologic therapy, investigational therapy or hormonal therapy within 14 days prior to the protocol-mandated 4-week drug holiday.
* Administration of any non-oncologic investigational drug within 30 days or five half-lives (whichever is longer) prior to the protocol-mandated 4-week drug holiday.
* Any ongoing toxicity from prior anti-cancer therapy that is > Grade 1 and/or that is progressing in severity, except alopecia.
* Known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to pazopanib or excipients that contraindicates participation.
* An untreated tumor growth rate of < 6.1% during the Screening period may exclude some patients.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2013-04; Primary Completion 2017-01 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
4-month Progression Free Survival (PFS) per RECIST version 1.1 guidelines | 4 months from the beginning of study treatment
  The primary objective of the study is to evaluate the 4-month PFS (with demonstrated increase in tumor doubling time) of eligible subjects treated with pazopanib according to RECIST version 1.1 guidelines.
  Tumor growth rate will be calculated by measuring growth at the specified intervals for the single, longest dimension of the tumor(s) (RECIST) and by calculating the area of the tumor(s), which will be the product of the longest dimension of the tumor(s) multiplied by its longest, perpendicular dimension (WHO).
  Progressive disease (PD) for target lesions is defined as at least a 20% increase in the sum of diameters of the target lesions taking as reference the smallest sum on study, and an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered progression.
  PD for non-target lesions is defined as unequivocal appearance of one or more new malignant lesions. Unequivocal progression of existing non-target lesions.

SECONDARY OUTCOMES:
4-month PFS per WHO criteria | 4 months from the beginning of study treatment
  The primary objective of the study is to evaluate the 4-month PFS (with demonstrated increase in tumor doubling time) of eligible subjects treated with pazopanib according to RECIST version 1.1 guidelines. The study statistician will calculate tumor growth rate per WHO criteria based on bidimensional tumor measurements (i.e., longest dimension of the tumor(s) and its longest perpendicular dimension) at each imaging time point.
Pharmacokinetics evaluation | Day 1 of Cycles 2 and 3 (Approximately 5 and 7 weeks from the start of study treatment)
  Evaluate the pharmacokinetics of pazopanib to define correlation of minimal drug concentrations with PFS, RR, duration of response, OS, and safety. Samples will be collected on Day 1 of Cycles 2 and 3 for plasma pazopanib trough PKs to assess the population of subjects with concentration greater than the target of 15 µg/mL.
Tumor growth kinetics | Assessed at Week -4 and 3 to 5 days prior to study treatment, approximately 4 weeks from the start of study treatment and every 6 weeks thereafter until the patient progresses or 60 months from the end of treatment, whichever occurs first
  Evaluate the tumor growth kinetics, both within subject, and across subjects over time and the change associated with pazopanib. Examine the correlation between tumor growth kinetics with pazopanib pharmacokinetics.
Response rate per RECIST version 1.1 | Assessed at Week -4 and 3 to 5 days prior to study treatment, approximately 4 weeks from the start of study treatment and every 6 weeks thereafter until the patient progresses or 60 months from the end of treatment, whichever occurs first
  Response rate (RR), where response is defined as complete response (CR) or partial response (PR) according to RECIST version 1.1 guidelines.
Overall Survival (OS) | Cycle 1 Day 1 (start of study treatment) up to death or 60 months after the end of study treatment, whichever occurs first
  The time origin for OS will be Cycle 1, Day 1. Subjects will be followed for up to 24 months after the end of treatment or until death, lost to follow-up, or withdrawal of consent, whichever occurs first.
PFS | Assessed at Week -4 and 3 to 5 days prior to study treatment, approximately 4 weeks from the start of study treatment and every 6 weeks thereafter until the patient progresses or 60 months from the end of treatment, whichever occurs first
  The time origin for PFS will be Cycle 1, Day 1. Repeat radiological imaging will be conducted after every 2 cycles of treatment (approximately 8 weeks)to evaluate disease status per RECIST v.1.1 and WHO criteria. Subjects who discontinue study treatment for reasons other than disease progression will continue to have their disease status reported every 3 months post end of treatment up to 60 months.
Response rate per WHO criteria | Assessed at Week -4 and 3 to 5 days prior to study treatment, approximately 4 weeks from the start of study treatment and every 6 weeks thereafter until the patient progresses or 60 months from the end of treatment, whichever occurs first
  Response rate (RR), where response is defined as complete response (CR) or partial response (PR) per WHO criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Warren A Chow, MD, Study Chair — City of Hope Medical Center
Locations (4):
- United States (4):
  - City of Hope, Duarte, California
  - Massachusetts General Hospital/Dana Farber Cancer Institute, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Frankel P, Ruel C, Uche A, Choy E, Okuno S, Somiah N, Chow WA. Pazopanib in Patients with Osteosarcoma Metastatic to the Lung: Phase 2 Study Results and the Lessons for Tumor Measurement. J Oncol. 2022 Jan 15;2022:3691025. doi: 10.1155/2022/3691025. eCollection 2022. PMID 35075361